CLINICAL TRIAL: NCT04336423
Title: Analysis of the Microbiome in the Healthy Smokers and COPD Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sei Won Lee, Division of Pulmonology and Critical Care Medicine, Department of Internal Medicine, University of Ulsan College of Medicine, Asan Medical Center, Seoul, South Korea, Asan Medical Center
Other Study IDs: Microbiome cohort
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Microbiota
Keywords: Chronic obstructive pulmonary disease; Microbiome
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Defecation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — sputum, fecal samples every 6 months for 30 healthy smokers for 3 years sputum, fecal samples every 3 months for 30 COPD patients for 3 years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy smoker: Healthy smokers with smoking history at least 10 pack-years and normal spirometry value
  Interventions: Diagnostic Test: Obtain samples from sputum and feces
- COPD patient: Patients with smoking history at least 10 pack-years and persistent airflow limitation that was not fully reversible (e.g. post-bronchodilator forced expiratory volume in 1 second/forced vital capacity (FEV1/FVC) <0.7)
  Interventions: Diagnostic Test: Obtain samples from sputum and feces

INTERVENTIONS:
Diagnostic Test: Obtain samples from sputum and feces — Samples are obtained from participants. No further intervention is required. Obtained samples will be further analyzed.

SUMMARY:
This study is to build a microbiome cohort by collecting sputum and fecal samples every few months for three years from healthy smokers and chronic obstructive pulmonary disease (COPD) patients. The aim of this study is to analyze the composition of microbiome of various samples (e.g. sputum, feces) and describe the difference between healthy smokers and COPD patients.

DETAILED DESCRIPTION:
After the introduction of the gut-lung axis theory, extensive studies revealed the diversity of microbiomes among healthy smokers and COPD patients form the respiratory samples or lung tissues. In the previous study, distinct difference in composition of microbiome in lung tissue between healthy smokers and COPD patients was reported. This study is to build a microbiome cohort by collecting sputum and fecal samples every few months for three years from healthy smokers and chronic obstructive pulmonary disease (COPD) patients who are being followed up by Asan Medical Center. The aim of this study is to analyze the composition of microbiome of various samples (e.g. sputum, feces) and describe the difference between healthy smokers and COPD patients. This study would help establishing gut-lung axis model in humans.

ELIGIBILITY:
Inclusion Criteria:

* Patients with smoking history at least 10 pack-year
* Patients with persistent airflow limitation that was not fully reversible (e.g. post-bronchodilator forced expiratory volume in 1 second/forced vital capacity (FEV1/FVC) <0.7)

Exclusion Criteria:

* Patients with co-existing illness that would interfere with study results (e.g., malignancy, congestive heart failure, cerebrovascular disorders, chronic renal failure, diabetes with severe complications, or uncontrolled hypertension)
* Patients with respiratory disease other than obstructive lung disease (e.g., previous pulmonary resection, tuberculosis-destroyed lung, and bronchiectasis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy smoker Healthy smokers with smoking history at least 10 pack-years and normal spirometry value
  COPD patient Patients with smoking history at least 10 pack-years and persistent airflow limitation that was not fully reversible (e.g. post-bronchodilator forced expiratory volume in 1 second/forced vital capacity (FEV1/FVC) <0.7)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-04-06 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Alpha diversity measured by operational taxonomic unit (OTU) quantitative analysis | An average of 3 months
  DNA is extracted from each sample from each patient by using a DNA Isolation Kit. The 16S universal primers are used for amplification of 16S ribosomal ribonucleic acid (rRNA) genes with polymerase chain reaction (PCR) system. After amplication, sequencing is performed using the GREENGENES database, after which a metagenomic analysis was performed by the MD Healthcare corporation using MDx-Pro software (Ver.1, Seoul, South Korea). Taxonomic assignment of these sequences is carried out with an operational taxonomic unit (OTU) cutoff of 3%.
Microbiome composition by metagenomic analysis | An average of 3 months
  The composition of microbiome is presented as bar graph.

SECONDARY OUTCOMES:
Biodiversity described by the Shannon diversity index and the Simpson index | An average of 3 months
  The Shannon index and the Simpson index is calculated by using metagenomic data.
Biodiversity described by Principal Component Analysis (PCA) | An average of 3 months
  PCA is performed for all 16S rRNA gene reads clustered at a 97% similarity.

CONTACTS AND LOCATIONS:
Overall Officials: Sei Won Lee, M.D. Ph.D., Principal Investigator — University of Ulsan College of Medicine, Asan Medical Center
Locations (1):
- Department of Pulmonary and Critical Care Medicine and Clinical Research Center for Chronic Obstructive Airway Diseases, Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erb-Downward JR, Thompson DL, Han MK, Freeman CM, McCloskey L, Schmidt LA, Young VB, Toews GB, Curtis JL, Sundaram B, Martinez FJ, Huffnagle GB. Analysis of the lung microbiome in the "healthy" smoker and in COPD. PLoS One. 2011 Feb 22;6(2):e16384. doi: 10.1371/journal.pone.0016384. PMID 21364979
- [Background] Kim HJ, Kim YS, Kim KH, Choi JP, Kim YK, Yun S, Sharma L, Dela Cruz CS, Lee JS, Oh YM, Lee SD, Lee SW. The microbiome of the lung and its extracellular vesicles in nonsmokers, healthy smokers and COPD patients. Exp Mol Med. 2017 Apr 14;49(4):e316. doi: 10.1038/emm.2017.7. PMID 28408748
- [Background] Morris A, Beck JM, Schloss PD, Campbell TB, Crothers K, Curtis JL, Flores SC, Fontenot AP, Ghedin E, Huang L, Jablonski K, Kleerup E, Lynch SV, Sodergren E, Twigg H, Young VB, Bassis CM, Venkataraman A, Schmidt TM, Weinstock GM; Lung HIV Microbiome Project. Comparison of the respiratory microbiome in healthy nonsmokers and smokers. Am J Respir Crit Care Med. 2013 May 15;187(10):1067-75. doi: 10.1164/rccm.201210-1913OC. PMID 23491408
- [Background] Cabrera-Rubio R, Garcia-Nunez M, Seto L, Anto JM, Moya A, Monso E, Mira A. Microbiome diversity in the bronchial tracts of patients with chronic obstructive pulmonary disease. J Clin Microbiol. 2012 Nov;50(11):3562-8. doi: 10.1128/JCM.00767-12. Epub 2012 Aug 22. PMID 22915614